CLINICAL TRIAL: NCT06013462
Title: DMEK Endothelial Keratoplasty in Patients With a History of Anterior or Posterior Segment Surgery : Serious Complication Rate and Visual Efficacy at 12 Months
Brief Title: DMEK Endothelial Keratoplasty in Patients With a History of Anterior or Posterior Segment Surgery
Acronym: DMEK complexes
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ASD_2023_6
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Patients Undergoing DMEK With a History of Anterior or Posterior Segment Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Descemet Membrane Endothelial Keratoplasty — DMEK (Descemet Membrane Endothelial Keratoplasty) is a surgical technique used to treat primary or secondary corneal endothelial decompensation.

SUMMARY:
DMEK (Descemet Membrane Endothelial Keratoplasty) is a surgical technique used to treat primary or secondary corneal endothelial decompensation. At the Rothschild Foundation, as in many Western referral centers, DMEK is currently the surgical technique of choice for the treatment of primary or secondary corneal endothelial decompensation.

Technically challenging, it is a relatively tedious surgery to learn, but offers the best visual and refractive results, as well as faster visual and functional recovery in simple cases.

In patients without anterior or posterior segment surgical history, the complication rate of DMEK, including graft rejection, is similar to that of other endothelial keratoplasty surgical techniques.

However, in specific cases, in patients with a history of ophthalmological surgery such as vitrectomy, trabeculectomy, large iris defects, anterior synechiae, aniridia or aphakia, the scientific literature shows a higher complication rate for DMEK (increased rate of rebulling and graft decompensation).

As a result, other techniques that are less effective on visual results continue to be used for these patients in a large number of centers.

Nonetheless, in our department, DMEK is also performed on these complicated patients.

When it comes to patients with a history of anterior or posterior segment surgery, it seems to us that the surgeons' experience with DMEK allows better visual results than with any other technique, but without any back up regarding the complication rate in the literature.

The main aim of this study is to describe, in patients with a history of anterior or posterior segment surgery undergoing DMEK, the 12-months occurrence rate of at least one serious post-operative complication.

ELIGIBILITY:
Inclusion Criteria :

* Patients scheduled for corneal endothelial transplantation in one or both eyes
* History of vitrectomy, trabeculectomy, large iris defects, anterior synechiae on the eye to be operated on
* Pseudophakia or aphakia in the eye to be operated on
* Express consent to participate in the study
* Affiliated or beneficiary of a social security scheme

Exclusion Criteria :

* Need for combined PKE + EK surgery
* Primary endothelial decompensation
* At least one contraindication to endothelial transplantation :

  * Presence of a stromal corneal cleft
  * Inflammatory or degenerative corneal pathology other than endothelial
  * Progressive corneal infection
  * Degenerative retinal pathology not allowing visual recovery postoperatively (for the purposes of this study, we accept patients who have had retinal detachment and whose loss of vision is clearly attributable to endothelial decompensation)
  * End-stage glaucoma not allowing visual recovery post-operatively (for this study, we accept patients who have had filtering surgery for glaucoma, which is stabilized at the time of surgery. Decline in vision must be clearly attributable to endothelial decompensation)
* Medical contraindication to general or local anesthesia
* Patient under legal protection
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group of 80 patients admitted for consultation at the Hôpital Fondation Adolphe de Rothschild up to one year prior to endothelial transplantation and meeting the above eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence rate of at least one serious DMEK post-op complication | 12 months
  Composite endpoint made of 4 serious post-op complications :
  * Rebulling : graft detachment of more than one-third of its surface area one week after surgery (on Avanti OCT-cornea), requiring air or gas injection in the anterior chamber.
  * Graft failure : no improvement in pachymetry at three months post-op (Avanti OCT-cornea).
  * Graft rejection : presence of cellular Tyndall in the anterior chamber and/or retro-descemetic precipitates and/or focal or diffuse increase in pachymetry > 20μm (Avanti OCT-cornea and slit-lamp biomicroscopic examination).
  * Macular cystoid edema : presence of intraretinal fluid in the macular area (macular OCT).

SECONDARY OUTCOMES:
Rebulling occurrence rate | 12 months
  Graft detachment of more than one-third of its surface area one week after surgery (on Avanti OCT-cornea), requiring air or gas injection in the anterior chamber.
Graft failure occurrence rate | 12 months
  No improvement in pachymetry at three months post-op (Avanti OCT-cornea).
Graft rejection occurrence rate | 12 months
  Presence of cellular Tyndall in the anterior chamber and/or retro-descemetic precipitates and/or focal or diffuse increase in pachymetry > 20μm (Avanti OCT-cornea and slit-lamp biomicroscopic examination).
Macular cystoid edema occurrence rate | 12 months
  Presence of intraretinal fluid in the macular area (macular OCT).
Intraocular hypertension occurrence rate | 12 months
  Intraocular pressure greater than 21mmHg measured by pneumotonometer or applanation tonometer.
Graft detachment (with or without rebulling) occurrence rate | 12 months
  Failure of the graft to press against the posterior host corneal stroma (Avanti OCT-cornea and slit-lamp biomicroscopic examination).
Surgeon's subjective assessment of surgical complexity | Right after the completion of the surgery
  Evaluation by the main surgeon at the end of the procedure, on a Likert scale from 0 to 10 (0 being normal, uncomplicated surgery and 10 being the maximum level of complexity encountered).
Duration of surgical procedure (in minutes) | Right after the completion of the surgery
  The start of the procedure is defined by the placement of the blepharostat and the end of the procedure is defined by the end of the lens dressing.
Evolution of visual results (corrected and uncorrected) | 1 month after surgery
  Measurements with optotypes :
  Best monocular visual acuity (decimal scale converted to logMAR)
Evolution of visual results (corrected and uncorrected) | 3 months after surgery
  Measurements with optotypes :
  Best monocular visual acuity (decimal scale converted to logMAR)
Evolution of visual results (corrected and uncorrected) | 6 months after surgery
  Measurements with optotypes :
  Best monocular visual acuity (decimal scale converted to logMAR)
Evolution of visual results (corrected and uncorrected) | 12 months after surgery
  Measurements with optotypes :
  Best monocular visual acuity (decimal scale converted to logMAR)
Evolution of refractive results | 1 month after surgery
  Nidek® autorefractometer measurement :
  1. Sphere (in dioptres)
  2. Cylinder (in dioptres)
  3. Spherical equivalent (in dioptres)
  4. Cylinder axis (in degrees)
Evolution of refractive results | 3 months after surgery
  Nidek® autorefractometer measurement :
  1. Sphere (in dioptres)
  2. Cylinder (in dioptres)
  3. Spherical equivalent (in dioptres)
  4. Cylinder axis (in degrees)
Evolution of refractive results | 6 months after surgery
  Nidek® autorefractometer measurement :
  1. Sphere (in dioptres)
  2. Cylinder (in dioptres)
  3. Spherical equivalent (in dioptres)
  4. Cylinder axis (in degrees)
Evolution of refractive results | 12 months after surgery
  Nidek® autorefractometer measurement :
  1. Sphere (in dioptres)
  2. Cylinder (in dioptres)
  3. Spherical equivalent (in dioptres)
  4. Cylinder axis (in degrees)
Evolution of endothelial loss | 1 month after surgery
  Measurement by central and peripheral specular microscopy (4 measurements performed nasally, temporally, superiorly and inferiorly). Endothelial loss in each quadrant is defined as a decrease in endothelial count (cells/mm²) expressed as a % relative to the pre-operative measurement.
Evolution of endothelial loss | 3 months after surgery
  Measurement by central and peripheral specular microscopy (4 measurements performed nasally, temporally, superiorly and inferiorly). Endothelial loss in each quadrant is defined as a decrease in endothelial count (cells/mm²) expressed as a % relative to the pre-operative measurement.
Evolution of endothelial loss | 6 months after surgery
  Measurement by central and peripheral specular microscopy (4 measurements performed nasally, temporally, superiorly and inferiorly). Endothelial loss in each quadrant is defined as a decrease in endothelial count (cells/mm²) expressed as a % relative to the pre-operative measurement.
Evolution of endothelial loss | 12 months after surgery
  Measurement by central and peripheral specular microscopy (4 measurements performed nasally, temporally, superiorly and inferiorly). Endothelial loss in each quadrant is defined as a decrease in endothelial count (cells/mm²) expressed as a % relative to the pre-operative measurement.
Evolution of corneal thickness | 1 month after surgery
  Corneal thickness in μm measured by OCT - Avanti® type cornea.
Evolution of corneal thickness | 3 months after surgery
  Corneal thickness in μm measured by OCT - Avanti® type cornea.
Evolution of corneal thickness | 6 months after surgery
  Corneal thickness in μm measured by OCT - Avanti® type cornea.
Evolution of corneal thickness | 12 months after surgery
  Corneal thickness in μm measured by OCT - Avanti® type cornea.
Evolution of posterior keratometry | 1 month after surgery
  Posterior keratometry in diopters measured by Scheimpflug corneal topography (Pentacam®).
Evolution of posterior keratometry | 3 months after surgery
  Posterior keratometry in diopters measured by Scheimpflug corneal topography (Pentacam®).
Evolution of posterior keratometry | 6 months after surgery
  Posterior keratometry in diopters measured by Scheimpflug corneal topography (Pentacam®).
Evolution of posterior keratometry | 12 months after surgery
  Posterior keratometry in diopters measured by Scheimpflug corneal topography (Pentacam®).

CONTACTS AND LOCATIONS:
Overall Officials: Alain SAAD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France